CLINICAL TRIAL: NCT06603805
Title: Optimal Surgical Approach for Early-Stage Breast Cancer in Chinese Patients Aged ≤ 40 Years: a Cohort Study
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Liu, Principal Investigator, West China Hospital
Other Study IDs: 2020427
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast-conserving surgery; radiotherapy; mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Radiotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MAST group: patients 1) aged between 18-40 years; 2) with a primary pathological diagnosis of invasive breast cancer; 3) receiving MAST; 4) having detailed information on T stage, N stage, clinical stage, hormone receptor status, endocrine therapy, and targeted therapy.
  Interventions: Procedure: MAST group
- BCS+RT group: Patients 1) aged between 18-40 years; 2) with a primary pathological diagnosis of invasive breast cancer; 3) receiving BCS+ RT; 4) having detailed information on T stage, N stage, clinical stage, hormone receptor status, endocrine therapy, and targeted therapy.
  Interventions: Procedure: breast-conserving surgery plus adjuvant radiotherapy

INTERVENTIONS:
Procedure: MAST group
  Groups: MAST group
Procedure: breast-conserving surgery plus adjuvant radiotherapy — Patients with early-stage (stage I, stage II, T≤2), and having the willingness to receive BCS were treated with BCS. All patients with BCS received post-surgery radiotherapy. Radiotherapy was administrated with a prescribed dose of 40 Gy in 15 fractions with photons and a boost of 10-16 Gy in 5-8 fractions with electrons to the ipsilateral breast. If axillary lymph nodes were involved, a conventional fraction was delivered with a prescribed dose of 50 Gy in 25 fractions to the ipsilateral breast and draining lymph node regions.
  Groups: BCS+RT group

SUMMARY:
The optimal surgical treatment option (BCS+RT versus MAST) for young patients with early-stage breast cancer remains debated. The present study aims to explore trends in surgical management and compare survival outcomes between BCS+RT and MAST in young patients with early-stage breast cancer, ultimately providing optimal treatment strategies for Asian populations.

DETAILED DESCRIPTION:
This study is a unique addition to the current research on young women with early-stage breast cancer, aiming to compare the survival outcomes between BCS+RT and MAST, providing valuable insights into their effectiveness for this group of patients. This study enrolled patients at West China Hospital, Sichuan University. Kaplan-Meier analyses with the log-rank test were applied to compare the locoregional recurrence-free survival (LRFS), distant metastasis-free survival (DMFS), breast cancer-specific survival (BCSS), and overall survival (OS). Cox multivariate hazard regression was employed to assess hazard ratios (HRs) between the two groups for survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 years.
* Pathological diagnosis of invasive breast cancer.
* Undergoing Breast-Conserving Surgery (BCS) with Radiotherapy (RT) or Mastectomy (MAST).
* Availability of detailed clinical information, including:

Tumor (T) stage. Node (N) stage. Clinical stage. Hormone receptor status. Endocrine therapy details. Targeted therapy details.

Exclusion Criteria:

* Male patients.
* Patients with distant metastatic disease.
* Patients with bilateral breast cancer.
* Patients not undergoing surgery.
* Follow-up time of less than 1 month.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patient data were extracted from the West China Hospital database at Sichuan University. Records between 1 January 2008 and 31 December 2019 were included.
Sampling Method: Non-Probability Sample
Enrollment: 974 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Breast cancer-specific survival (BCSS) | Jan 1, 2008 to 31 Dec, 2019
LRFS (Locoregional Recurrence-Free Survival) | Jan 1, 2008 to 31 Dec, 2019
DMFS (Distant Metastasis-Free Survival) | Jan 1, 2008 to 31 Dec, 2019
OS (Overall Survival) | Jan 1, 2008 to 31 Dec, 2019

IPD SHARING:
Plan to Share IPD: Undecided